CLINICAL TRIAL: NCT05098626
Title: Investigation of Spinal Health and Internet Addiction of Individuals Working Remotely
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aybüke Fanuscu, Research Assistant, Hacettepe University
Other Study IDs: HUSpine013
Record Dates: First submitted 2021-10-16; First posted 2021-10-28 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Posture; Spine; Internet Addiction; Neck Pain; Low Back Pain
Keywords: Posture; Spine; Neck pain; Low back pain; Screen time; Internet addiction
MeSH Terms: conditions — Internet Addiction Disorder; Neck Pain; Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals Working Remotely: Individuals aged between 18-60 and working remotely, who volunteered to participate in the study, will form the study group.

SUMMARY:
Low back pain and neck pain are common problems that affect people at certain times in their lives. These people constitute a significant part of the disease burden due to their recurrent complaints. People with low back and neck pain often seek medical attention. This situation causes individuals to apply to the hospital frequently and causes a serious cost at the social level.

When the risk factors for neck pain are examined, many factors such as genetics, sleep problems, smoking, obesity, sedentary lifestyle, poor posture, previous neck pain, trauma, back pain and poor general health cause neck pain to develop. Similarly, conditions such as age, obesity, and poor general health appear to be risk factors for low back pain. In addition to these risk factors, it has been reported that occupational factors such as long and sedentary working hours and unsuitable workplace conditions may also cause low back and neck pain. Fixed posture and prolonged sitting are thought to be risk factors for low back and neck pain, but opinions on this subject are not clear.

The COVID-19 pandemic has created a global crisis since 2019 and caused a change in the lifestyle of all people around the world. The World Health Organization (WHO) stated that social distance should be increased and face-to-face contact should be reduced to prevent the spread of the pandemic. For this reason, many institutions have decided to work remotely and trainings have been carried out remotely. The increasing teleworking style with the COVID-19 pandemic has led to an increase in the average screen time of individuals. It was reported that time spent on the Internet increased by 52% compared to the pre-pandemic period.

This study aims to investigate the relationship between increased teleworking hours and internet use during the pandemic period in individuals with low back or neck pain. Researchers think that postural changes that may occur with increased distance working time, increased fixed posture and asymmetrical loading may contribute to the uncertain relationship between low back and neck pain and posture.

ELIGIBILITY:
Inclusion Criteria:

* Working online during the pandemic process,
* Have a smart phone,
* Agree to voluntarily participate in the research.

Exclusion Criteria:

* Have a malignant condition,
* Loss of function due to neurological or systemic disease,
* Having had a surgical operation in the last 6 months,
* Have an unhealed fracture,
* Withdraw consent at any stage of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals working remotely during the pandemic
Sampling Method: Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2022-03-20 (Estimated); Primary Completion 2022-06-20 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Craniovertebral Angle | 5 minutes, in one assessment session.
  Global Postural System (GPS) will be used for posture evaluation. GPS is a computerized photographic postural assessment system. It consists of a digital camera, a ruler frame, and a stable platform that allows for consistent landmark identification. The craniovertebral angle will be recorded, which provides the most relevant and reproducible data in the assessment of neck posture with GPS. The craniovertebral angle is the angle between a line drawn between the C7 vertebra and the tragus and a horizontal line drawn from C7
Evaluation of Sternocleidomastoideus Muscle Architecture | 5 minutes, in one assessment session.
  Sternocleidomastoideus muscle will be architecturally evaluated by US using a 5-12 MHz linear probe (GE Logiq E5 ultrasound device) at rest and during muscle activation. Muscle thickness and pennation angle will be recorded.
Evaluation of Internet Addiction | 10 minutes, in one assessment session.
  This evaluation will be carried out using the Kimberly Young Internet Addiction Questionnaire. The questionnaire consisting of 20 items; evaluate their dependencies in personal, professional and social functions. The questions are scored between 0 and 5 points. A total score between 0 and 30 indicates a normal level of internet use, total scores between 31 and 49 indicate the presence of mild addiction, a total score between 50 and 79 indicates the presence of a moderate level of addiction, and a total score of over 80 indicates the presence of severe internet addiction.

SECONDARY OUTCOMES:
Evaluation of the Time Spent in Front of the Screen | 2 minutes, in one assessment session.
  he time spent in front of the screen will be evaluated by questioning the average time spent by people on three different devices as computer, tablet and phone use.
Evaluation of Body Mass Index | 2 minutes, in one assessment session.
  Body Mass Index (BMI), muscular and fat body weights will be assessed with TANITA BC420SMA (Tanita Corp, Tokyo, Japan). TANITA is a medically approved and reliable measuring device. It determines body composition by taking advantage of changes in bioelectrical resistance.
Evaluation of Low Back Disability | 5 minutes, in one assessment session.
  It was developed to evaluate the level of functional loss in individuals with low back pain. The scale consists of 10 questions about pain intensity, self-care, lifting-carrying, walking, sitting, standing, sleep, degree of change in pain, travel and social life. Each question is scored between 0-5 points. The total score is evaluated out of 100. A high score means an increased level of disability.
Evaluation of Neck Disability | 5 minutes, in one assessment session.
  The Neck Disability Questionnaire includes a total of 10 questions about pain, personal care, concentration, work, driving, and sleeping. Each question is scored between 0-5 points. 0-4 points means no disability, 5-14 points means mild disability, 15-24 points means moderate disability, 25-34 points means severe disability, 35 points and above means complete disability. The total score is evaluated out of 50.

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin Özel Aslıyüce, MSc, Study Chair — Hacettepe University; Dilara Onan, MSc, Study Chair — Hacettepe University; Müzeyyen Öz, MSc, Study Chair — Hacettepe University; Özlem Ülger, Professor, Study Director — Hacettepe University

IPD SHARING:
Plan to Share IPD: No